CLINICAL TRIAL: NCT06345872
Title: SPIN Opioid: Improving Sleep and Reducing Opioid Use in Individuals With Chronic Pain
Brief Title: Improving Sleep and Reducing Opioid Use in Individuals With Chronic Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY005883; 1R01DA054311 (NIH)
Record Dates: First submitted 2024-03-28; First posted 2024-04-03 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Chronic Pain; Chronic Insomnia; Opioid Use
Keywords: Chronic pain; Chronic insomnia; Opioid use; CBT-I
MeSH Terms: conditions — Chronic Pain; Sleep Initiation and Maintenance Disorders | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): 8 weeks of online CBT-I (1 session/week for 1 hour), followed by tapered withdrawal and motivational interviewing and check-ins.
  Interventions: Behavioral: CBT-I; Other: Tapered Withdrawal
- Treatment as usual (Other): Continuation of standard treatment for sleep and pain for 8 weeks, followed by tapered withdrawal and motivational interviewing and check-ins.
  Interventions: Behavioral: Treatment as usual; Other: Tapered Withdrawal

INTERVENTIONS:
Behavioral: CBT-I — Includes 8 weekly sessions of CBT-I and 2 bi-monthly boosters. Each session is to be completed individually by the participant in a single sitting (less than 45 mins). Each session should be completed in 7 days with next session released only after prior one completed.
  Arms: Experimental
Behavioral: Treatment as usual — Includes 8 weekly sessions of standard treatment and 2 bi-monthly boosters. Each session is to be completed individually by the participant in a single sitting (less than 45 mins). Each session should be completed in 7 days with next session released only after prior one completed.
  Arms: Treatment as usual
Other: Tapered Withdrawal — Individualized gradual tapered withdrawal following CDC guidelines, additional check-ins and motivational interviewing with a therapist.

SUMMARY:
The goal of this study is to test two behavioral interventions for chronic insomnia in individuals with chronic pain and use prescribed opioid medication to treat their chronic pain.

DETAILED DESCRIPTION:
Opioid therapy is commonly prescribed for patients with chronic widespread musculoskeletal pain, but offers questionable benefit for long-term pain management and is associated with arrhythmias, overdose, and death. Individuals with chronic pain experience high rates of comorbid chronic insomnia, arousal, and abnormal brain activation in response to painful stimuli. Research shows individuals with chronic pain exhibit increased brain activation in regions associated with pain modulation in response to painful stimuli compared to healthy controls. Withdrawal from opioids is difficult; and inadequately managed pain contributes to that difficulty. The Cognitive Activation Theory of Stress (CATS) tests the hypothesis that poor sleep and arousal lead to critical changes in brain activation that increase pain severity and lead to opioid use. Research shows cognitive behavioral treatment for insomnia (CBT-I, an evidence based intervention for chronic insomnia) improves sleep, arousal, abnormal brain activation, and pain in individuals with comorbid chronic pain and insomnia, but does not reduce opioid use. However, because CBT-I improves each of the mediators hypothesized to contribute to opioid use, it warrants examination as a neoadjuvant to gradual tapering of opioid medication. The proposed trial tests the novel hypothesis that improving sleep and decreasing arousal will lead to normalized brain activation and decreased pain prior to gradual tapering, which will facilitate reduced opioid use. This hypothesis is supported by theory (CATS) and empirical findings. It also reflects federal pain research priorities.

ELIGIBILITY:
Inclusion Criteria:

* 18+ yrs
* willing to be randomized,
* can read/understand English
* diagnosed with chronic widespread pain and insomnia (as described below)
* prescribed opioid medication for 1+ mo, 3+ times per week
* desire to reduce or eliminate opioid use
* written agreement from physician prescribing opioid medication
* no prescribed or OTC sleep meds for 1+ mo, or stabilized on meds for 6+ wks

Exclusion Criteria:

* unable to provide informed consent
* cognitive impairment (MMSE <26)
* sleep disorder other than insomnia [i.e., sleep apnea (apnea/hypopnea index, AHI >15)
* Periodic Limb Movement Disorder (myoclonus arousals per hour >15)]
* bipolar or seizure disorder (due to risk of sleep restriction treatment)
* other severe, untreated major psychopathology except for depression or anxiety (e.g.,suicidal ideation/intent, psychotic disorders)
* psychotropic or other medications (e.g., beta-blockers) that alter pain or sleep (medications prescribed for pain or sleep are allowed)
* participation in other non-pharmacological treatment for pain, sleep, or mood outside the current trial
* internal metal objects or electrical devices
* pregnancy
* presumptive/confirmed lumbar nerve root compression
* confirmed lumbar spinal stenosis
* <6 mos post-back surgery
* other spinal disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 165 (Estimated)
Dates: Start 2024-12-11 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Change in Insomnia Severity Index | Single administration at baseline, 8 weeks, following completion of gradual tapered withdrawal, and 6 month follow-up
  Insomnia severity; score range 0-28 (low severity - high severity)
Change in Pain Intensity - Daily Electronic Sleep Diaries | Single administration at baseline, 8 weeks, following completion of gradual tapered withdrawal, and 6 month follow-up
  Daily electronic dairies will record pain unpleasantness; range: 0-100 (none- most unpleasantness)
Change in Wake After Sleep Onset - Daily Electronic Sleep Diaries | Single administration at baseline, 8 weeks, following completion of gradual tapered withdrawal, and 6 month follow-up
  Daily electronic dairies will record wake after sleep onset (number of minutes)
Change in Sleep Onset Latency- Daily Electronic Sleep Diaries | Single administration at baseline, 8 weeks, following completion of gradual tapered withdrawal, and 6 month follow-up
  Daily electronic dairies will record sleep onset latency (number of minutes)
Change in Sleep Efficiency- Daily Electronic Sleep Diaries | Single administration at baseline, 8 weeks, following completion of gradual tapered withdrawal, and 6 month follow-up
  Daily electronic dairies will record sleep efficiency
Change in Fatigue - Daily Electronic Sleep Diaries | Single administration at baseline, 8 weeks, following completion of gradual tapered withdrawal, and 6 month follow-up
  Daily electronic dairies will record insomnia severity; range: 0-100 (no insomnia - most severe)
Change in Sleep and Pain Medication - Daily Electronic Sleep Diaries | Single administration at baseline, 8 weeks, following completion of gradual tapered withdrawal, and 6 month follow-up
  Daily electronic dairies will record daily medication consumption)
Change in Perceived Stress Scale | Single administration at baseline, 8 weeks, following completion of gradual tapered withdrawal, and 6 month follow-up
  Perception of stress; score range: 0-40 (low stress - high stress)
Change in Peripheral Arousal | 5 mins at rest at baseline, 8 weeks, following completion of gradual tapered withdrawal, and 6 month follow-up
  Heart Rate Variability (as measured by Holter-Monitoring)
Change in Neural Imaging: Structural/Functional MRI/Diffusion Weighted Imaging | Single administration at baseline, 8 weeks, following completion of gradual tapered withdrawal, and 6 month follow-up
  Assessment of neural plasticity
Change in Thermal Pain Response | Single administration at baseline, 8 weeks, following completion of gradual tapered withdrawal, and 6 month follow-up
  Participants will undergo quantitative sensory testing using a contact thermode applied to the left plantar, VAS scale for pain ()-100)
Change in Opioid Use (Quantitative) | Single administration at baseline, 8 weeks, following completion of gradual tapered withdrawal, and 6 month follow-up
  Change in opioid use assessed with quantitative urine opioid panel
Change in Opioid Use (Self-Report) | Single administration at baseline, 8 weeks, following completion of gradual tapered withdrawal, and 6 month follow-up
  Change in opioid use assessed with daily electronic diaries

SECONDARY OUTCOMES:
Change in Objective Wake After Sleep Onset (Actigraph) | Single administration at baseline, 8 weeks, following completion of gradual tapered withdrawal, and 6 month follow-up
  Wake after sleep onset via GENEActiv
Change in Objective Sleep Onset Latency (Actigraph) | Single administration at baseline, 8 weeks, following completion of gradual tapered withdrawal, and 6 month follow-up
  Sleep Onset Latency via GENEActiv
Change in Objective Sleep Efficiency (Actigraph) | Single administration at baseline, 8 weeks, following completion of gradual tapered withdrawal, and 6 month follow-up
  Sleep Efficiency via GENEActiv
Change in Neural Connectivity: Structural/Functional MRI/Diffusion Weighted Imaging | Single administration at baseline, 8 weeks, following completion of gradual tapered withdrawal, and 6 month follow-up
  Assessment of brain connectivity
Short Inventory of Problems | Single administration at baseline, 8 weeks, following completion of gradual tapered withdrawal, and 6 month follow-up
  Modified from validated alcohol survey for opioid related problems
Change in Pain Catastrophizing Scale | Single administration at baseline, 8 weeks, following completion of gradual tapered withdrawal, and 6 month follow-up
  The PCS yields a total score and three subscale scores assessing rumination, magnification and helplessness. Total score range from 0-52, with higher scores indicating greater pain catastrophizing.

OTHER OUTCOMES:
Change in 36-Item Short Form Survey (SF-36) | Single administration at baseline, 8 weeks, following completion of gradual tapered withdrawal, and 6 month follow-up
  Self-reported health; score range: low quality of life to high quality of life
Change in Depression (Beck Depression Inventory-II) | Single administration at baseline, 8 weeks, following completion of gradual tapered withdrawal, and 6 month follow-up
  Depression severity; score range: 0-63 (normal - extreme depression)
Change in State-Trait Anxiety Inventory (STAI) | Single administration at baseline, 8 weeks, following completion of gradual tapered withdrawal, and 6 month follow-up
  Trait and state anxiety; score range: 20-80 (low anxiety - high anxiety)
Medications/Substances Uses and Dosages | Single administration at baseline, 8 weeks, following completion of gradual tapered withdrawal, and 6 month follow-up
  Non-opioid pain/sleep medication use and dosage, tobacco, caffeine, alcohol, marijuana via daily electronic diaries
Change in Subjective Opioid Withdrawal Scale (SOWS) | Single administration at 8 weeks, following completion of gradual tapered withdrawal, and 6 month follow-up
  Monitor changes in withdrawal symptoms
Change in Opioid Cravings Scale | Single administration at baseline, 8 weeks, following completion of gradual tapered withdrawal, and 6 month follow-up
  Monitor of cravings related to opioid use
Change in NIH Toolbox | Single administration at baseline, 8 weeks, following completion of gradual tapered withdrawal, and 6 month follow-up
  20-minute of two computerized cognitive tasks

CONTACTS AND LOCATIONS:
Overall Officials: Christina S McCrae, PhD, Principal Investigator — University of South Florida; Britani Holland, PhD, Study Director — University of South Florida
Locations (1):
- University of South Florida, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McCrae CS, Williams J, Roditi D, Anderson R, Mundt JM, Miller MB, Curtis AF, Waxenberg LB, Staud R, Berry RB, Robinson ME. Cognitive behavioral treatments for insomnia and pain in adults with comorbid chronic insomnia and fibromyalgia: clinical outcomes from the SPIN randomized controlled trial. Sleep. 2019 Mar 1;42(3):zsy234. doi: 10.1093/sleep/zsy234. PMID 30496533
- [Background] McCrae CS, Curtis AF, Miller MB, Nair N, Rathinakumar H, Davenport M, Berry JR, McGovney K, Staud R, Berry R, Robinson M. Effect of cognitive behavioural therapy on sleep and opioid medication use in adults with fibromyalgia and insomnia. J Sleep Res. 2020 Dec;29(6):e13020. doi: 10.1111/jsr.13020. Epub 2020 Mar 3. PMID 32126156
- [Background] Morin CM, LeBlanc M, Daley M, Gregoire JP, Merette C. Epidemiology of insomnia: prevalence, self-help treatments, consultations, and determinants of help-seeking behaviors. Sleep Med. 2006 Mar;7(2):123-30. doi: 10.1016/j.sleep.2005.08.008. Epub 2006 Feb 3. PMID 16459140
- [Background] McCrae CS, Mundt JM, Curtis AF, Craggs JG, O'Shea AM, Staud R, Berry RB, Perlstein WM, Robinson ME. Gray Matter Changes Following Cognitive Behavioral Therapy for Patients With Comorbid Fibromyalgia and Insomnia: A Pilot Study. J Clin Sleep Med. 2018 Sep 15;14(9):1595-1603. doi: 10.5664/jcsm.7344. PMID 30176973
- [Background] Seal KH, Shi Y, Cohen G, Cohen BE, Maguen S, Krebs EE, Neylan TC. Association of mental health disorders with prescription opioids and high-risk opioid use in US veterans of Iraq and Afghanistan. JAMA. 2012 Mar 7;307(9):940-7. doi: 10.1001/jama.2012.234. PMID 22396516
- [Background] Martinez MP, Miro E, Sanchez AI, Diaz-Piedra C, Caliz R, Vlaeyen JW, Buela-Casal G. Cognitive-behavioral therapy for insomnia and sleep hygiene in fibromyalgia: a randomized controlled trial. J Behav Med. 2014 Aug;37(4):683-97. doi: 10.1007/s10865-013-9520-y. Epub 2013 Jun 7. PMID 23744045